CLINICAL TRIAL: NCT05416307
Title: A Multipart, Open-label, Single-arm, Multicenter Study to Evaluate the Safety, Efficacy and Pharmacokinetics of ELA026 in Participants With Secondary Hemophagocytic Lymphohistiocytosis (sHLH)
Brief Title: Open-label Study of ELA026 in Participants With Secondary Hemophagocytic Lymphohistiocytosis (sHLH)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Electra Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ELA026-CP002
Record Dates: First submitted 2022-06-06; First posted 2022-06-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Secondary Hemophagocytic Lymphohistiocytosis (sHLH)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 ELA026 (Experimental): Cohort 1: Single dose escalation up to 3.0 mg/kg IV or SC.
  Cohort 2: priming dose: 0.1 mg/kg IV on Day 1; 0.3 mg/kg IV on Day 2 - 4, followed by weekly maintenance doses of 1 mg/kg IV/SC from Day 8 to Day 81.
  Cohort 3: priming dose: 0.1 mg/kg IV on Day 1; 0.3 mg/kg IV on Days 2 - 4, followed by twice weekly maintenance doses of 0.5 mg/kg IV/SC from Day 8 to Day 81.
  Interventions: Drug: ELA026
- Part 2 ELA026 (Experimental): Cohort A and Cohort B: priming dose: 0.1 mg/kg IV on Day 1; loading dose 0.3 mg/kg IV on Days 2- 4, followed by twice weekly maintenance doses of 0.5 mg/kg (IV/SC) from Day 8 to Day 81.
  Interventions: Drug: ELA026

INTERVENTIONS:
Drug: ELA026 — Multiple doses of ELA026

SUMMARY:
Hemophagocytic lymphohistiocytosis is a rare, aggressive and life-threatening syndrome of excessive immune activation. Secondary hemophagocytic lymphohistiocytosis (sHLH) is the most common form of this disease and is typically associated with several other clinical conditions (eg, malignancy associated HLH (mHLH), infection, or autoimmune disease). ELA026 is a fully human immunoglobulin G1 (IgG1) signal regulatory protein (SIRP)-directed monoclonal antibody designed to deplete the myeloid and T cells driving the inflammation. The purpose of this study is to assess the safety, efficacy pharmacokinetics and pharmacodynamics of ELA026 in participants with sHLH.

DETAILED DESCRIPTION:
This study consists of two parts: Phase 1b (Part 1) and Phase 2/3 (Part 2).

Part 1 is designed to evaluate the safety, efficacy, pharmacodynamics, and pharmacokinetics of ELA026 in pediatric and adult participants with treatment-naïve (TN) and relapsed/refractory sHLH. The main objectives of Part 1 are to determine the safety of ELA026 administered intravenously (IV) and subcutaneously (SC) to participants with sHLH and to identify the recommended Phase 3 dose and schedule for ELA026. Participants will be enrolled into a dose-escalating cohort (Cohort 1) followed by two fixed dose cohorts (Cohorts 2-3) treated over 12-weeks.

Part 2 (SURPASS) is designed as an open-label, single-arm, multicenter, historical control registrational study to evaluate ELA026 in newly diagnosed TN adult and pediatric sHLH participants. All participants are diagnosed with HLH-2004 criteria unless indicated. Cohort A (primary cohort) will enroll newly diagnosed TN participants ≥18 years old with mHLH. Cohort B (exploratory cohort) will enroll participants including ≥18 years old participants with TN sHLH not triggered by malignancy; ≥18 years old participants with newly diagnosed TN mHLH diagnosed by biomarker criteria but not meeting HLH-2004 diagnostic criteria; and 6 to 17 year old participants with newly diagnosed TN sHLH (due to any trigger). For 6 to 12 year old participants, there is a safety lead-in cohort with refractory sHLH.

Part 1 is closed to recruitment and Part 2 is recruiting for eligible participants.

ELIGIBILITY:
Key Inclusion Criteria for Part 1:

1. ≥12 years at the time of HLH diagnosis (Cohort 1).
2. ≥6 years at the time of HLH diagnosis (Cohort 2-3).
3. Treatment naïve or relapsed/refractory (Cohorts 1 and 2).
4. Treatment naïve or early refractory (Cohort 3).
5. Participant with sHLH confirmed criteria based on fulﬁlling 5 out of 8 HLH-2004 diagnostic criteria.

Key Inclusion Criteria for Part 2:

1. Cohort A: Adults with newly diagnosed, treatment-naïve, malignancy-associated sHLH.
2. Cohort B: Adults with newly diagnosed, treatment-naïve, non-malignancy-associated sHLH.
3. Cohort B: Adults with newly diagnosed, treatment-naïve, malignancy-associated sHLH, diagnosed by OHI index.
4. Cohort B: 13 to 17 years olds with newly diagnosed, treatment-naïve sHLH.
5. Cohort B: 6 to 12 year olds, with refractory sHLH (safety lead-in cohort).
6. Cohort B: 6 to 12 year olds, with newly diagnosed, treatment-naïve sHLH (after completion of safety lead-in cohort).

Key Exclusion Criteria for Part 1:

1. Known or previous treatment for primary HLH
2. Any other significant concurrent, uncontrolled medical condition that in the opinion of the Investigator contraindicates participation in this study
3. Unknown trigger for sHLH
4. Active, relapsed/refractory malignancy for which no suitable therapies are available to treat the malignancy triggering the HLH
5. Allogeneic hemopoietic stem cell transplant (HSCT) within 100 days of the first dose of ELA026.
6. Ongoing administration of any therapies used to treat HLH (excluding dexamethasone)
7. Live or attenuated vaccine received within 6 weeks or bacille Calmette-Guerin (BCG) vaccine within 12 weeks prior to Screening

Key Exclusion Criteria for Part 2:

1. Refractory sHLH (except for the safety lead-in cohort for 6-12 year olds in Cohort B).
2. Known or suspected primary or hereditary HLH.
3. Severe organ dysfunction.
4. Any other signiﬁcant concurrent, uncontrolled medical condition that contraindicates participation in this study or prohibits completion of study procedures.
5. End-stage malignancy for which no suitable therapies are available to treat the malignancy triggering the HLH.
6. Allogeneic hemopoietic stem cell transplant within 100 days prior to the first dose of ELA026.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participant with Incidence of Treatment-Emergent Adverse Events (TEAEs) [Safety and tolerability] | Up to Week 12
  Incidence of adverse events (AEs) including dose-limiting toxicities (DLTs), serious adverse events (SAEs), deaths, AEs leading to withdrawal from study
Part 2 (Cohort A): 56-day Survival Rate in Participants with mHLH and Have Lymphoma as the Cancer Trigger | 56 days

SECONDARY OUTCOMES:
Number of Participants Achieving Early Survival (Cohort A) | up to 90 days
Number of Participants Achieving HLH Disease Response by Day 29 (Cohort A) | Up to Day 29
  HLH disease response includes achievement of CR, mCR, PR, or HI.
Number of Participants with TEAEs | Up to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Electra Therapeutics Inc.
Locations (34):
- United States (14):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California, Los Angeles, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Columbia University, New York, New York
  - Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Germany (2):
  - Universitätsklinikum Jena, Jena, Thuringia
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen, Villingen-Schwenningen
- Italy (5):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - Bambino Gesu' Roma, Roma
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Materno-Infantile Burlo Garofolo, Trieste
- Netherlands (3):
  - Amsterdam Universitair Medische Centra - Locatie Academisch Medisch Centrum, Amsterdam, Noord-Holland - NET
  - Erasmus UMC, Rotterdam
  - Wilhelmina Kinderziekenhuis, Utrecht
- Spain (7):
  - Clinica Universidad de Navarra - Madrid, Madrid, Madrid - SPA
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre - SPA
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla - SPA
  - Hospital Universitari i Politecnic La Fe, Valencia, Valencia - SPA
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital La Fe Valencia, Valencia
- University College London Hospitals NHS Foundation Trust, London, England - UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No